CLINICAL TRIAL: NCT06007703
Title: Evaluation of the Safety and Effectiveness of the Global Treatment Including Multilayer Compression Therapy (Urgo KTwo®) in Addition to an Interactive Dressing (UrgoStart® Plus) in the Management of Venous Leg Ulcers
Brief Title: Evaluation of the Efficacy of Multilayer Compression & UrgoStart Plus
Status: Completed | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23/003/GHT; 327680 (Other: South West - Cornwall & Plymouth Research Ethics Committee)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcer; Venous Ulcer; Venous Insufficiency of Leg; Leg Ulcer
Keywords: Ulcer; Venous
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, venous leg ulcers have been very difficult to manage, with associated poor healing rates, and the likelihood of recurrence. Even following correction of underlying venous dysfunction, ulcers can take time to respond to conventional treatment with compression therapy. Recently, the leg ulcer service in Gloucestershire - part of the vascular surgical team - have been using an interactive dressing called UrgoStart Plus under compression therapy in the management of chronic venous leg ulcers and we have experienced some positive outcomes for otherwise recalcitrant ulcers.

A previous study published in 2017 by Meaume et al demonstrated a reduction in wound surface area after 8 weeks of treatment with UrgoStart Plus. However, whether or not use of the dressing, in combination with compression bandages, improves 12-week healing rates, remains an unanswered question.

The aim of the proposed study is to provide an evaluation of this interactive dressing when used under compression bandages and to compare 12-week healing rates with a similar cohort of patients who have been treated with a simple low adherent dressing under compression. This has been our gold standard up to now and we have been collecting prospective data from patients treated in our unit.

DETAILED DESCRIPTION:
Leg ulcers are notoriously difficult to treat with poor outcomes often reported. The majority of these ulcers are caused by a deficient venous return from the to lower leg and the mainstay in treatment is compression therapy and further venous treatments such as foam sclerotherapy. However, some ulcers still take many months to heal causing great suffering and reduced quality of life and great expense to the NHS.

More knowledge has been gained concerning the impact of protease (enzyme) activity in venous leg ulcers and high numbers of these could contribute to the non-healing state. UrgoStart Plus is an interactive dressing which has a protease modulating effect and has been shown to reduce proteases and improve healing. The CHALLENGE trial published by Meaume et al (2012) showed significant reductions in wound surface area following eight weeks of treatment with UrgoStart for venous leg ulcers and diabetic foot ulcer. However, there is no published data as yet evaluating impact on healing of venous ulcers at 12 weeks.

The present study aim is to evaluate the 12-week healing rates in patients with venous leg ulcers treated in a proven compression system using UrgoStart Plus as the wound contact layer. This can be compared with 12-week healing for a similar cohort of patients treated with the same compression system and a simple low adherent non-interactive dressing.

ELIGIBILITY:
Inclusion Criteria:

* Related to the patient:
* Patient over 18 years old who has provided his/her written informed consent,
* Patient who is able and willing to commit to regular follow up with the investigating team for the purpose of the study, and in line with established service protocols for routine patient follow up until ulcer healed,
* Patient who agrees to adhere to the study protocol with respect to the type of multilayer compression system and primary wound dressing,

Related to the venous leg ulcer:

* Ulcer between 2 and 20 cm² in surface,
* Ulcer duration less than six weeks ("new ulcer"),
* Venous leg ulcer - Ankle Brachial Pressure Index > 0.85 at baseline, done in the previous three months and if not, at the inclusion of the patient),

Exclusion Criteria:

Related to the patient:

* Patient participating in another clinical trial,
* Patient with known hypersensitivity to one of the components of the tested compression system Urgo KTwo Lite Latex free or the UrgoStart dressings,
* Patient who is unable to tolerate compression therapy,
* Patient presenting a neoplastic lesion treated by radiotherapy or chemotherapy or patients treated with immunosuppressive drugs or high-dose corticosteroids,
* Patient with a history of deep or superficial vein thrombosis in the 3 months prior to inclusion,
* Patient confined to bed.

Related to the leg ulcer:

* Ulcer with ABPI<0.85,
* Ulcer which is clinically infected,
* Ulcer surface area partially or totally covered by black necrosis plaque,
* Malignant ulcer,
* Ulcer less than 3 cm, from any edge, to another wound located on the same limb.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients recruited for this clinical investigation will be patients treated on an outpatient basis for a venous leg ulcer presenting with an ABPI>0.85 (venous origin). This is in accordance with local management protocol.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Time to healing | 12 weeks
  Complete ulcer closure (100% re-epithelialisation) after a maximum of 12 weeks treatment period.

SECONDARY OUTCOMES:
Patient health related quality of life | 12 weeks
  Patient Quality of Life through a specific Wound Quality of Life Questionnaire testing 17 aspects of the leg ulcer and how it impacts on the participant with scores from 0-4 for each statement. The higher the score, the worse the impact.

CONTACTS AND LOCATIONS:
Overall Officials: Colin E Davies, MSc, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Gloucestershire Royal Hospital, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meaume S, Truchetet F, Cambazard F, Lok C, Debure C, Dalac S, Lazareth I, Sigal ML, Sauvadet A, Bohbot S, Dompmartin A; CHALLENGE Study Group. A randomized, controlled, double-blind prospective trial with a Lipido-Colloid Technology-Nano-OligoSaccharide Factor wound dressing in the local management of venous leg ulcers. Wound Repair Regen. 2012 Jul-Aug;20(4):500-11. doi: 10.1111/j.1524-475X.2012.00797.x. Epub 2012 Jun 8. PMID 22681551

DOCUMENTS (2):
  • Study Protocol (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT06007703/Prot_000.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT06007703/ICF_001.pdf